CLINICAL TRIAL: NCT00856271
Title: A Randomized, Double-blind, Double-dummy, Multi-center Study to Investigate the Safety and Efficacy of Olmesartan Medoxomil Compared With Losartan Potassium in Patients With Mild to Moderate Essential Hypertension
Brief Title: Olmesartan Medoxomil Versus Losartan Potassium in Patients With Mild to Moderate Essential Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Collaborators: Shanghai Sankyo Pharmaceuticals Co., Ltd. (Unknown)
Responsible Party: Naotaka Ikegami, Vice President, Shanghai Sankyo Pharmaceuticals, Co., Ltd.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SS-866/01
Record Dates: First submitted 2009-03-03; First posted 2009-03-05 (Estimated); Last update posted 2010-09-29 (Estimated); Status verified 2010-09

CONDITIONS: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension | interventions — Olmesartan Medoxomil; Losartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): olmesartan medoxomil
  Interventions: Drug: olmesartan medoxomil
- 2 (Active Comparator): losartan potassium
  Interventions: Drug: losartan potassium

INTERVENTIONS:
Drug: olmesartan medoxomil — oral tablets, once daily for 8 weeks
  Arms: 1
Drug: losartan potassium — capsules, once daily for 8 weeks
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of olmesartan medoxomil compared with losartan potassium in patients with mild to moderate essential hypertension.

ELIGIBILITY:
Inclusion Criteria:

* mild to moderated essential hypertension (mean seated diastolic blood pressure ≥ 95 mmHg and <110 mmHg, mean seated systolic blood pressure < 180 mmHg)
* able to give written informed consent

Exclusion Criteria:

* known or suspected secondary hypertension
* history of chronic hepatic diseases
* obstructive hypertrophic cardiomyopathy/clinically significant valvular heart disease
* cardiac arrhythmia
* unstable angina pectoris
* congestive heart insufficiency (New York Heart Association classification III-IV)
* bilateral renal artery stenosis
* isolated renal artery stenosis
* post renal transplantation
* history of acute myocardial infarction/percutaneous transluminal coronary angioplasty or heart surgery within three months before enrollment
* retina bleeding/effusion
* insulin dependent diabetes mellitus
* uncontrolled non-insulin dependent diabetes mellitus

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 287 (Actual)
Dates: Start 2004-08; Primary Completion 2005-02 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Change of trough seated diastolic blood pressure from baseline to 8 weeks | Baseline to 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Vice President, Study Director — Sankyo Shanghai Pharmaceuticals
Locations (5):
- China (5):
  - Beijing
  - Chongqing
  - Guangzhou
  - Nanjing
  - Shanghai